CLINICAL TRIAL: NCT01566149
Title: An Open-Label Study to Assess the Safety and Tolerability of Zenhale® (a Fixed-Dose Combination of Mometasone Furoate/Formoterol Fumarate Delivered by Metered Dose Inhaler) in 40 Subjects With Persistent Asthma (Protocol No. 206-00 [P08212])
Brief Title: Study of Mometasone Furoate/Formoterol Fumarate (MF/F) Metered Dose Inhaler (MDI) in Adolescents & Adults With Persistent Asthma (P08212)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08212; MK-0887A-206 (Other: Merck Study ID)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Formoterol Fumarate; Mometasone Furoate, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MF/F 200/10 mcg MDI BID (Active Comparator): Participants receiving MF/F 200/10 mcg MDI twice daily (BID) for 12 weeks
  Interventions: Drug: Mometasone Furoate/Formoterol Fumarate (MF/F) 100/5 mcg MDI
- MF/F 400/10 mcg MDI BID (Active Comparator): Participants receiving MF/F 400/10 mcg MDI BID for 12 weeks
  Interventions: Drug: Mometasone Furoate/Formoterol Fumarate (MF/F) 200/5 mcg MDI

INTERVENTIONS:
Drug: Mometasone Furoate/Formoterol Fumarate (MF/F) 100/5 mcg MDI — Two oral inhalations per dose
  Other Names: Zenhale®; SCH 418131; MK-0887A
  Arms: MF/F 200/10 mcg MDI BID
Drug: Mometasone Furoate/Formoterol Fumarate (MF/F) 200/5 mcg MDI — Two oral inhalations per dose
  Other Names: Zenhale®; SCH 418131; MK-0887A
  Arms: MF/F 400/10 mcg MDI BID

SUMMARY:
The purpose of this study is to assess the safety, tolerability & effectiveness of 2 strengths of Mometasone Furoate/Formoterol Fumarate (MF/F) Metered Dose Inhaler (MDI) in the treatment of persistent asthma in adults & adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma of at least 6 months duration
* Current use of a medium or high daily dose of an inhaled corticosteroid (ICS) (alone or in combination with a long-acting beta agonist [LABA]) for at least 6 weeks prior to Screening AND must be on a stable asthma regimen (daily dose unchanged) for at least 2 weeks prior to Screening
* Agrees to change asthma therapy (if changing asthma therapy poses no inherent risk)
* If female of reproductive potential, agrees to remain abstinent or use 2 acceptable methods of birth control during study participation. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy, hormonal contraceptive

Exclusion Criteria:

* Treatment in the emergency room (for a severe asthma exacerbation), or admitted to the hospital for management of airway obstruction within previous 3 months
* Any prior ventilator support for respiratory failure secondary to asthma,
* Upper or lower respiratory tract infection (viral or bacterial) within previous 2 weeks
* History of a medical condition that, in the investigator's opinion, may interfere with study participation,
* History of smoking within previous year or a cumulative smoking history of more than 10 pack-years
* Known allergy to or intolerance of ICSs, LABAs, or any of the ingredients included in the study medications
* History of use of illicit drugs
* Inability to correctly use an oral MDI
* Pregnant, breastfeeding or plans to become pregnant during study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one study site in Vietnam between March 2012 and September 2012.
Pre-assignment Details: Participants who were previously on medium-dose asthma medication were assigned to Mometasone Furoate/Formoterol Fumarate (MF/F) 200/10 mcg Metered Dose Inhaler (MDI) twice daily (BID) and participants who were previously on high-dose asthma medication were assigned to MF/F 400/10 mcg MDI BID.
Groups:
- MF/F 200/10 mcg MDI BID: Participants receiving MF/F 200/10 mcg MDI BID for 12 weeks
Period: Overall Study
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Started | 24 | 25
Completed | 21 | 23
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Non-compliance with study medication | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (14.48) | 41.2 (14.91) | 38.3 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least One Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Up to Week 14
Population: The Full Analysis Set (FAS) population consisted of all participants assigned treatment who received at lease one dose of study medication.
Measure: Number; unit: participants
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Number analyzed (Participants) | 24 | 25
participants | 5 | 8

2. Primary Outcome: Number of Participants With At Least One Drug-Related AE
Description: A drug-related AE was defined as any AE for which there is reasonable possibility of drug relationship as assessed by the Investigator.
Time Frame: Up to Week 14
Population: The FAS population consisted of all participants assigned treatment who received at lease one dose of study medication.
Measure: Number; unit: participants
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Number analyzed (Participants) | 24 | 25
participants | 0 | 0

3. Primary Outcome: Number of Participants With At Least One Serious AE
Description: A serious AE was defined as any untoward medical occurrence or effect that at
  any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly or birth defect; and/or cancer.
Time Frame: Up to Week 14
Population: The FAS population consisted of all participants assigned treatment who received at lease one dose of study medication.
Measure: Number; unit: participants
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Number analyzed (Participants) | 24 | 25
participants | 0 | 0

4. Primary Outcome: Number of Participants Who Discontinued From the Study Due to an AE
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Up to Week 12
Population: The FAS population consisted of all participants assigned treatment who received at lease one dose of study medication.
Measure: Number; unit: participants
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Number analyzed (Participants) | 24 | 25
participants | 0 | 1

5. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: Baseline was defined as the highest FEV1 value of three assessments prior to first dose of study drug. If two (or all three) spirometry efforts had identical FEV1, the FEV1 from the effort with the highest Forced Vital Capacity (FVC) was to be recorded. Week 12 FEV1 was assessed as the morning FEV1 at the end of the dosing interval (trough FEV1). For participants who discontinued prior to Week 12, the FEV1 measurement from the discontinuation visit was to be be carried forward to Week 12 if (and only if) the participant's study medication compliance rate prior to discontinuation was at least 85%.
Time Frame: Baseline and Week 12
Population: The FAS population consisted of all participants assigned treatment who received at lease one dose of study medication and had at least one efficacy measurement post-dose.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Number analyzed (Participants) | 24 | 25
liters
  Baseline FEV1 | 2.397 (0.6824) [0.006 to 0.214] | 2.215 (0.6206) [-0.051 to 0.153]
  Week 12 FEV1 | 2.503 (0.7418) | 2.270 (0.6041)
  Change from Baseline in FEV1 at Week 12 | 0.106 (0.2892) | 0.054 (0.2055)

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: The FAS population consisted of all participants assigned treatment who received at least one dose of study medication.
Arm/Group | MF/F 200/10 mcg MDI BID | MF/F 400/10 mcg MDI BID
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 5/24 | 8/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F 200/10 mcg MDI BID (N=24) | MF/F 400/10 mcg MDI BID (N=25)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.